Unique Protocol ID: 2014/7951

Secondary Ids: 2014/878 [Regional Committee for Medical Research Ethics Norway]

# Pediatric Pain Management Practices in Postoperative Units – an Intervention Study

## Research Group

- Anja Hetland Smeland, Pediatric Nurse, MSc, PhD student, Children's Surgical Department, Oslo University Hospital
- Tone Rustøen, RN, PhD, Researcher, Division of Emergencies and Critical Care, Department of Research and Development, Oslo University Hospital and Professor II, Department of Nursing Science, University of Oslo (supervisor)
- Alison Twycross, PhD, DMS, CertEd(HE), RGN, RMN, RSCN, Editor in Evidence Based Nursing and Reader in Children's Pain Management, Head of Department for Children's Nursing, Department of Children's Nursing Faculty of Health and Social Care, London South Bank University (co- supervisor)
- Stefan Lundeberg MD, PhD, Senior Consultant, Pain Treatment Service, Astrid Lindgren Children's Hospital, Stockholm (Intervention study)
- Hanne Reinertsen, Associate Professor, Oslo and Akershus University college of applied Sciences (Intervention study)
- Lill Nybro, MSc student, Intensive Care Nurse, Oslo University Hospital (interview with children)
- Torgun Næss, MSc student, Pediatric Nurse, Oslo University Hospital (interview with children)
- Eva Carlsen, Pediatric Nurse, Children's Surgical Department, Oslo University Hospital (facilitator Intervention study)

# **Summary**

Despite available research on pediatric pain management, pain is still underestimated and undertreated. According to research, nurses' attitudes and lack of knowledge are some possible causes. This study will explore nurses' pediatric postoperative pain management practices. The aim is to evaluate if a tailored educational intervention with nurses working in postoperative units improve their knowledge and attitudes of pain management and pain management practices. This is a tailored educational intervention study with a pre-post design and a comparison group (baseline T-1, one month after intervention T-2, and six months after intervention T-3), including a sample of nurses working in six postoperative units. The units are the largest pediatric postoperative units of each of the six university hospitals, covering all health regions in Norway. Three different approches will be used (survey with questionnaire of the nurses, observations of clinical practice, and interviews with children) to collect data about pediatric pain management practices in this study.

Unique Protocol ID: 2014/7951

Secondary Ids: 2014/878 [Regional Committee for Medical Research Ethics Norway]

# **Background**

Pain in children and adolescents is underestimated and undertreated even if a lot of research is done in the area (1, 2). Research suggests that lack of knowledge about pain and pain management in children are one of the reasons for the undertreatment (3-14).

As late as in the 1970's and 80's premature and newborn children went through surgery without pain medication (15) because it was claimed that the children could not feel pain since the nervous system was not fully developed. More recent studies show that preterm infants are hypersensitive to pain (16), and that surgery in the neonatal period can lead to prolonged pain and hypersensitivity in the damaged area (17, 18).

Untreated pain can cause unnecessary suffering, increased risk of complications, increased risk of morbidity and mortality, as well as lead to longer hospital stays and increased cost (19). Long-term consequences of inadequate relief of acute pain can be chronic pain for 10-50% of the patients, of which 2-10% of them will experience severe chronic pain (19).

Nurses who work at postoperative units have a considerable responsibility to ensure optimal pain management. Research shows that the use of guidelines and pain assessment tools improve the pain treatment of children through systematic assessment and evaluation (20, 11). However, more than half of European hospitals are reported to lack written guidelines for pain treatment and more than half of the patients experience severe pain (21, 22).

Pain assessment in children is largely based on patients' self-reports and nurses' assessment and the use of observational pain assessment tools (23, 24). There are many types of pain assessment tools for children (behavior form, face form, numerical scales) (11, 25-29), but no pain assessment tools are suitable for all children as it must be selected on the basis of the child's age, developmental level and context (27).

Few studies have examined the effectiveness of educational interventions on pediatric nurses' pain management (7, 30-33). The studies showed improved perception of pain assessment and management (30), improved knowledge of pain management (7, 31,32) and increased use of non-pharmacological interventions (31). Johnston et al. (31) & Le May et al. (32) studied if there where any change in nurses' analgesic administration and found that there were no significant change. Vincent et al. (33) conducted a pilot intervention study which showed significant improvement in nurses' beliefs and pain management practices. All studies have small samples, except Ellis et al. (30), and only Johnston et al. (31) had a comparison group. None of these studies have measured if tailored educational intervention improve nurses' pediatric pain management practice by observing the nurses or examined the children's experience of pain and pain management. There is a need to explore this further.

# **Objectives**

The main objective of the present study is to improve pediatric postoperative pain management. This will be achieved by first exploring the pediatric postoperative pain management practice using different approaches (study 1). Then, an intervention will be developed based on the results from the first study and available research in the area (study 2). After that, we will investigate if the tailored interventions with nurses at postoperative units improve the nurses' knowledge of pediatric pain management and pediatric pain management practice (study 3). The different studies are presented in Table 1:

Table 1: The studies

| | Studies | Activity |
|---|---|---|
| Study 1 | Explore nurses' pediatric | Data collection (baseline T-1) using: |
| | postoperative pain practices | Questionnaire PNKAS-N |

Unique Protocol ID: 2014/7951

Secondary Ids: 2014/878 [Regional Committee for Medical Research Ethics Norway]

| | | Observational study of clinical practice |
|---|---|---|
| | | Interview with children |
| Study 2 | Develope a tailored educational intervention | Develope tailored educational intervention based on: |
| Study 3 | Implementation and evaluation of the intervention | Implementation of the intervention |

# **Study 1 Exploring Nurses' Pediatric Postoperative Pain Practices**

#### Research questions

What kind of knowledge and attitudes do nurses working in postoperative units have about pediatric pain management?

How do nurses manage the pediatric pain practices in postoperative units? What is the children's experience of pain and pain management after surgery?

Three different approches will be used (questionnaire, observation and interview) to collect data about pediatric pain management practices in this study.

# a) Survey with Questionnaires

Sample/Setting

The study will be conducted by nurses at six postoperative units, which have children and adolescents after surgery. The units are the largest pediatric postoperative units of each of the six university hospitals, covering all health regions in Norway. All nurses (259 nurses) working with patients in these units will be asked to participate in this study.

#### Data Collection

Data from the nurses regarding knowledge and attitudes toward pain management will be collected using "The Pediatric Nurses' Knowledge and Attitudes Survey Regarding Pain Questionnaire - Norwegian version" (PNKAS-N). The PNKAS was developed by Manworren (9) and translated into Norwegian tested and validated according to Norwegian conditions by Hovde et al. (5). The questionnaire is based upon guidelines for acute pain management in infants, children and adolescents, American Pain Society, The World Health Organization and the Joint Commission on Accreditation of Healthcare Organizations (9, 10). The PNKAS-N consist of 40 questions about general pain management, pain assessment, and use of pharmacological and non-pharmacological treatment of pain in children. Several items are related to areas in pediatric pain management where lack of knowledge has been reported. An appendix of the questionnaire register the nurses' age, education level, work experience and full-time equivalent. An additional section has been added to the questionnaire in order to get the staff views about the facilitators and barriers to optimized pain management. The PNKAS-

Unique Protocol ID: 2014/7951

Secondary Ids: 2014/878 [Regional Committee for Medical Research Ethics Norway]

N will be distributed to the nurses three times, at baseline (before the intervention), and one and six months after the intervention.

# Data Analysis

The data will be analyzed using statistical methods (SPSS). Descriptive and correlational statistics will be used to describe and summarize data (34, 35). Means, standard deviations, medians, and interquartile ranges will be calculated for continuous data. Frequency counts and proportions will be calculated for categorical data.

#### **b)** Observational Study

The aim of this part is to obtain more knowledge about how nurses actually manage postoperative pain in children and whether pain management practices adhere to current best practice guidelines.

#### Sample

Non-participant observational studies will be conducted at all six units at baseline. Each unit have 40-60 nurses working with patients and 10-15 children undergoing surgery every day, 50-75 children/week in total.

#### Data Collection

During each data collection period, observations will be carried out for four-hour periods (day and evening), two weeks per unit (40 hours per unit per occasion, 240 hours in total). The observational study will focus on observing the nurses general pain management practice, pain assessment (use of pain assessment tools), use of pharmacological and non-pharmacological treatment of pain in children. A checklist and field notes will be used based on the PNKAS-N themes and essential areas of pediatric pain management identified in a literature review (36). Field notes will include descriptions of what is occurring during the period of observation and records of comments made by nurses related to pediatric pain management. The field notes will be recorded partly during the observation and partly after the observation (directly after), depending on the situation at the unit. No data about the child will be recorded except age, gender, type of surgery, and days since surgery. The other data that will be recorded is what the situation gives, but no data that can identify the patient will be recorded. The checklist will be pilot tested based on two different observation situations.

# Data Analysis

Data from each nurse will be collected by using the pain management checklist and summarizing each of the nurses' pain management practices. A content analysis will be carried out on data within the field notes (37, 38). Information in the field notes will be examined for common themes (35, 39). Using highlighter pens, the researcher will code the data in each of the categories. After the data in the field notes are coded, the researcher will identify recurring themes and compare this to the data from the pain checklists to provide a picture of current pain management practices. The data will be given to another experienced pediatric nurse who will code the data without any knowledge of the themes identified by the researcher, to minimize researcher bias. After having coded the data the researcher and the second coder will discuss and agree upon the final wording of the themes.

# c) Interview with Children

The aim of this part is to obtain more knowledge about what are the children's experiences of pain and pain management after surgery.

Unique Protocol ID: 2014/7951

Secondary Ids: 2014/878 [Regional Committee for Medical Research Ethics Norway]

#### Sample

Twenty children older than six years going through surgery at the time of data collection at two of six units (randomly chosen), and their parents, will be asked to participate in this study.

#### Data Collection

The draw and write technique (40, 41, 42) will be adapted for use with children aged 6-9 years allowing them to draw and tell, draw and write or write their story about how well their pain has been managed in hospital. Older children will be offered the option of individual interviews. The semi-structured interview schedule will reflect the questions used by Polkki et al. (43) and the Royal College of Nursing (44) and include questions related to:

- Have you had any pain while you were in hospital?
- Were you asked if you had any pain?
- Who asked you about your pain?
- How did the nurses help you when you were in pain?
- Do you think nurses can help children in pain in a better way?
- What is tolerable pain to you?
- Do you have pain at rest and when you move?
- Does the pain limit your daily activities?

All children will be asked to rate the worst pain experienced during the first 48–72 hours postoperatively using a numeric rating scale (NRS) from 0 "no pain" to 10 "worst pain imaginable" or a face scale depending on their cognitive capabilities. All children taking part in the study will also be asked to rate the worst pain experienced during the post-operative period as well as their current level of pain. These interviews will take place before the child is discharged from hospital, and all interviews will be tape recorded. The interview guide will be pilottested in two different interviews.

# Data Analysis

Children's responses to the interview questions will be transcribed verbatim. Content analysis will be used to analyse the transcripts using a five-step approach (45):

- 1 Creating and organising files for data
- 2 Reading through the text and forming initial codes
- 3 Describing the social setting, people involved and events
- 4 Analysing data for identifying emerging themes
- 5 Interpreting and making sense of the findings

# **Study 2 Develop the Tailored Educational Intervention**

The intervention will be developed based on available research, results from baseline in the present study and staff views about the facilitators and barriers to optimized pediatric pain management of the included units.

The intervention will be a one day seminar for nurses working at the units, with lectures and workshops with main focus on the subjects showing the lowest pediatric pain management competence. In addition, there will be clinical supervision in pediatric postoperative pain management (two or three days per unit). The intervention will be conducted by two experts (nurse and physician) in pediatric postoperative pain management.

Unique Protocol ID: 2014/7951

Secondary Ids: 2014/878 [Regional Committee for Medical Research Ethics Norway]

After the intervention there will be different reminders every week for the first month, and then every month (in different forms) about pediatric pain management during six months of time.

# Study 3 Implementation and Evaluation of the Intervention

# **Research Questions**

Will tailored educational interventions improve nurses' knowledge and attitude to pediatric pain management?

Will tailored educational intervention improve nurses' pediatric pain management practice?

After the educational intervention is implemented there will be different reminders. The first month there will be reminders every week, and thereafter every month for six months period of time. The reminders are based on the general pain management practice, pain assessment, pharmacological and non-pharmacological treatment of pain in children with main focus on the subjects showing the lowest pediatric pain management competence at baseline. The reminders will be in different forms (poster, pamphlet, picture, pocket guide etc.) posted in different places at the units (46).

After the intervention there will be an evaluation of the effectivness of intervention. To evaluate the intervention three different approches will be used (questionnaire, observation and interview) to collect data about pediatric pain management practices.

Pre-post tailored educational intervention design, with comparison group, measured during three periods; T-1 (baseline - before intervention), T-2 (one month after intervention) and T-3 (six months after intervention).

Table 2: FLOWCHARTS

# 

**Flowchart** 

Unique Protocol ID: 2014/7951

Secondary Ids: 2014/878 [Regional Committee for Medical Research Ethics Norway]

Three of these six units will be randomized (cluster randomized by units) in an intervention group and three in a comparison group. Each unit has about 40-60 nurses, approximately 260 nurses in total.

#### Data Collection

All nurses at all six units are asked to take part in the study by completing the PNKAS-N questionnaire at T-2 and T-3. Non-participant observational studies will be conducted at four units at T-2. Futhermore, one unit from the intervention group and one unit from the comparison group will be randomly chosen for observational studies at T-3. During each data collection period observations will be carried out for four-hour periods, two weeks per unit (40 hours per unit per occasions, 240 hours in total). Children older than six years who are having surgery at the time of data collection at the same two units will be asked to participate in an interview (20 children from two units) at T-2.

#### Data Analysis

Descriptive and inferential statistics will be used to analyse quantitative data at each data collection. Regression analyses that accounts for repeated measurements and cluster correlations (within units) will be used for comparisons between data collected at baseline T-1, T-2 and T-3. Content analysis will be used to analyse the children's responses to the interview questions. Supplementary data from the interviews and the observation studies at T-1 and T-2 will be compared to see if the tailored educational intervention improve nurses' pediatric pain management practice and childrens experience of pain assessment (e.g. use of pain assessment tools, use of pharmacological and non-pharmacological treatment of pain).

#### **Ethics:**

Ethical research guidelines will be followed (47-52). An approval from the Norwegian Social Science Data Services (NSD) and Regional Committee for Medical Research Ethics (REK South-East) will be obtained. Necessary approval from the hospitals will be obtained. Contact will be established with relevant persons at the units and cooperation on the implementation of the project. The project will be personally presented by the project manager at the relevant departments at baseline. A pilot observational study and two pilot interviews with children will be done before baseline (T-1).

Participants (nurses, children and their parents) will receive oral and written information about the study, and informed consents will be obtained from all the participants. The information letter includes information about the study, and explains that it is voluntary to participate in the study and the participants' answers will be treated anonymously (53-57).

The questionnaires will be distributed to the nurses with an information letter and an envelope for returning the questionnaires. Informed consents will be obtained from all the persons (nurses, children and their parents) who are present during the observational studies. The participants who do not approve will be excluded from the study. Informed consents will be obtained from both the children (> 12 years) and the parents that are participating in the interviews. All data will be recorded on standardized forms. The interviews with children will be coded so that no data collected include date of birth or other sensitive information that can identify the child. Data will be stored securely and deleted at the end of the study (58-61).

#### Benefit/Risk:

Participating in the study will involve some extra work in filling in the questionnaire and to participate in the intervention. Furthermore, the participants may feel uncomfortable being observed during the observational study. They will be informed that no data about any nurses

Unique Protocol ID: 2014/7951

Secondary Ids: 2014/878 [Regional Committee for Medical Research Ethics Norway]

or others will be avalaiable for others. It will also be voluntary to participate. Furthermore, the questionnaires are anonymous. Studying the nurses' knowledge and attitudes to pain in children and adolescents in Norway may lead to increased focus, awareness and attention on the topic among nurses. This means that while taking part in the study will not be of direct benefit to the children participating it may result in improved care for children in the future, The study will summarize Norwegian nurses' knowledge and attitudes to pain in children and adolescents. Further, the study will summarize nurses' use of pain assessment tools and if there are guidelines for pain assessment and treatment of the various units in the all health regions in Norway. The evaluation of the intervention can contribute to development of a national educational program for nurses in relation to post-operative pain and pain management in children and adolescents.

# **Declaration of Conflicting Interests:**

There are no conflicts of interest.

#### Schedule 2014-2019

| Schedule 2014-2019 | | | |
|---|---|---|---|
| Preparation | | November 2013 - June 2014 | |
| D ( 11 () | T. 1 | G 4 1 N 1 2014 | PNKAS-N<br>Observation |
| Data collection | T-1 | September - November 2014 | Interview with children |
| | intervention | January – February 2015 | |
| | | | PNKAS-N<br>Observation |
| | T-2 | March - April 2015 | Interview with children |
| | T-3 | September- October 2015 | PNKAS-N<br>Observastion |
| Data analysis | 1 3 | September 2015 - March 2017 | Coservasiion |
| Papers | paper 1 | December 2015 – March 2017 | |
| | paper 2 | April 2016 - March 2017 | |
| | paper 3 | October 2016 - November 2017 | |
| | paper 4 | October 2016 - November 2017 | |

# **Publication Plan:**

| | Nurses knowledge about pediatric postoperative pain management |
|---|---|
| | Data from baseline, PNKAS, observasjon (short summari in table) baseline |
| | Journal: Pain Management Nursing |
| | http://www.painmanagementnursing.org/content/authorinfo |
| | (Nurses' pediatric pain management practices in postoperative units in Norway |
| 2016 | - data will be from the questionnaires at baseline and the observation studies. ) |
| | Pain in children after surgery- an interview study |
| | Data from T1 |
| | Journal: Journal of Clinical Nursing |
| 2016 | http://onlinelibrary.wiley.com/journal/10.1111/(ISSN)1365-2702/homepage/ForAuthors.html |
| | The development of a tailored intervention about pediatric pain management after surgery |
| | (Data from baseline interview, baseline observation, PNKAS) |
| | Theoretical framework |
| 2017 | Journal: Scandinavian Journal of Caring Sciences |

Unique Protocol ID: 2014/7951

Secondary Ids: 2014/878 [Regional Committee for Medical Research Ethics Norway]

| | http://onlinelibrary.wiley.com/journal/10.1111/(ISSN)1471-6712/homepage/ForAuthors.html |
|---|---|
| | (A tailored educational intervention with nurses in pediatric pain management |
| | - the content of the intervention will be published were all the details will be given. ) |
| | Implementation and evaluation of an intervention about pediatric pain management after |
| | surgery |
| | Data: Endring fra T1, T2, T3- PNKAS, interview |
| | Journal: Pain |
| | http://edmgr.ovid.com/pain/accounts/ifauth.htm |
| | (Evaluation of a tailored educational intervention with nurses pediatric pain management |
| | - the main paper will describe the effect of the intervention. Data from all measurement points will be |
| 2017 | presented, and data from the interviews and observations will be given as well.) |

Even if only three publications will be included in the doctoral thesis, the reseach group will write the fourth one.

The results from the study will be presented at national as well as international conferences.

# **Dissemination of the results:**

| | | | National conference Norway |
|---|---|---|---|
| | | | NOSF, Oslo |
| Presentation | Oral | January 2017 | http://www.norsksmerteforening.no/kurs |
| | | | National conference Norway |
| | | | Norsk Barnesmerteforenings vårseminar, Oslo |
| Presentation | Oral | March 2017 | http://www.norskbarnesmerteforening.no/arrangementer |
| | | | National conference Norway |
| | | | BSF Vårseminar, Bergen |
| | | | http://www.reiseogkonferanseservice.com/Barnesykepleie |
| Presentation | Oral | April 2017 | rforbundet/Varseminar2017/program.cfm |
| | | | International Conference |
| | | | 11th International Symposium on Pediatric Pain (ISPP) |
| | | | Kuala Lumpur, Malaysia |
| Presentation | Poster | July 2017 | http://www.ispp2017.org/abstract |

Unique Protocol ID: 2014/7951

Secondary Ids: 2014/878 [Regional Committee for Medical Research Ethics Norway]

#### References

- 1 Hauer, J., Jones, B.L. & Wolfe, J., Poplack, D. G., Kim, M. S. (2015). Evaluation and management of pain in children. *UpToDate*. <a href="http://www.uptodate.com/contents/evaluation-and-management-of-pain-in-children?source=search">http://www.uptodate.com/contents/evaluation-and-management-of-pain-in-children?source=search</a> result&search=PAIN+CHILDREN&selectedTitle=1%7E150
- 2 IASP (2011c). Acute Pain management in Newborn Infants Pain. [Online]. <a href="http://www.iasp-pain.org/PublicationsNews/NewsletterIssue.aspx?ItemNumber=2075">http://www.iasp-pain.org/PublicationsNews/NewsletterIssue.aspx?ItemNumber=2075</a> & <a href="http://iasp.files.cms-plus.com/Content/ContentFolders/Publications2/PainClinicalUpdates/Archives/PCU\_19-6\_final\_12-8-11\_1390260191290\_1.pdf">http://www.iasp-pain.org/PublicationsNews/NewsletterIssue.aspx?ItemNumber=2075</a> & <a href="http://www.iasp-pain.org/Publications2/PainClinicalUpdates/Archives/PCU\_19-6\_final\_12-8-11\_1390260191290\_1.pdf</a>
- 3 Bernadi, M., Catania, G. & Tridello, G. (2007). Knowledge and attitudes about cancer pain management: a national survey of Italian hospice nurses. *Cancer Nurs*, 30(2), E20-6.
- 4 Coulling, S. (2005). Nurses' and doctors' knowledge of pain after surgery. Nurs Stand, 19(34), 41-49.
- 5 Hovde, K. R., Granheim, T. H., Christophersen, K.-A. & Dihle, A. (2012). The Norwegian Version of the Pediatric Nurses' Knowledge and attitudes Survey Regarding Pain: Reliability and Validity, *Pedatric nursing*, 38 (5), 264-269.
- 6 Hossain, S. (2010). Nurses' Knowledge and Attitudes, and Pain Management Practice of Post-Operative Children in Bangladesh. Prince of Songkla University. Nedlastet fra <a href="http://kb.psu.ac.th/psukb/bitstream/2010/7826/1/325999.pdf">http://kb.psu.ac.th/psukb/bitstream/2010/7826/1/325999.pdf</a>
- 7 Huth, M. M., Gregg, T. L., Lin, L. (2010). Education changes Mexican nurses' knowledge and attitudes regarding pediatric pain. *Pain Manag Nurs*. Dec;11(4):201-8. doi: 10.1016/j.pmn.2009.11.001.
- 8 Lewthwaite, B. J., Jabusch, K. M., Wheeler, B. J. Schnell-Hoehn, K. N., Mills, J., Estrella-Holder, E., Fedorowicz, A. (2011). Nurses' knowledge and attitudes regarding pain management in hospitalized adults. *J Contin Educ Nurs*, 42(6), 251-7. doi: 10.3928/00220124-20110103-03. Epub 2011 Jan 10. <a href="http://www.ncbi.nlm.nih.gov/pubmed/21229930">http://www.ncbi.nlm.nih.gov/pubmed/21229930</a>
- 9 Manworren, R.C. (2000). Pediatric nurses' knowledge and attitudes survey regarding pain. Pediatr Nurs, 26, 610-614. <a href="http://www.ncbi.nlm.nih.gov/pubmed/12026363">http://www.ncbi.nlm.nih.gov/pubmed/12026363</a>
- 10 Rieman, M. T., Gordon, M. & Marvin, J. M. (2007). Pediatric nurses' knowledge and attitudes survey regarding pain: a competency tool modification. *Pediatr Nurs*, 33, 303-306. http://www.ncbi.nlm.nih.gov/pubmed/17907730
- 11 Simons, J.M. & MacDonald, L.M. (2004). Pain assessment tools: children's nurses' views. *Journal of Child Health Care*, 8, 264. Doi: 10.1177/1367493504047317.
- 12 Twycross, A. (2007). What is the impact of theoretical knowledge on children's nurses' post-operative pain management practices? an exploratory study. *Nurse Educ Today*, 27, 697-707. <a href="http://www.ncbi.nlm.nih.gov/pubmed/17134793">http://www.ncbi.nlm.nih.gov/pubmed/17134793</a>
- 13 Smart, S. (2005). POST-OPERATIVE PAIN MANAGEMENT KNOWLEDGE AND ATTITUDES OF PAEDIATRIC NURSES:- A NEW ZEALAND REGIONAL VIEW. Victoria University of Wellington. [Online]. Tilgjengelig på <a href="http://researcharchive.vuw.ac.nz/bitstream/handle/10063/38/thesis.pdf?sequence=2">http://researcharchive.vuw.ac.nz/bitstream/handle/10063/38/thesis.pdf?sequence=2</a> [Lastet 13.april 2014]. <a href="http://researcharchive.vuw.ac.nz/handle/10063/38">http://researcharchive.vuw.ac.nz/handle/10063/38</a>
- 14 Vincent, C. V.H. (2005). Nurses' knowledge, attitudes, and practices: regarding children's pain. MCN Am J Matern Child Nurs, 30, 177-183.
- 15 Olsson, G., Jylli, L. (2001). Smärta hos barn och ungdomar. Lund, Sverige: Studentlitteratur.
- 16 Peters, J. W., Schouw, R., Anand, K. J. van Dijk, M., Duivenvoorden, H. J., Tibboel, D. (2005). Does neonatal surgery lead to increased pain sensitivity in later childhood? *Pain*, 114(3), 444-54.
- 17 Anand, K. J. S., Gracia-Preats, J. A. & Kim, M. S. (2015). Assessment of neonatal pain. *UpToDate*. <a href="http://www.uptodate.com/contents/assessment-of-neonatal-pain">http://www.uptodate.com/contents/assessment-of-neonatal-pain</a>
- 18 Anand, K. J. S., Gracia-Preats, J. A. & Kim, M. S. (2015). Prevention and treatment of neonatal pain. *UpToDate*. <a href="http://www.uptodate.com/contents/prevention-and-treatment-of-neonatal-pain?source=related\_link">http://www.uptodate.com/contents/prevention-and-treatment-of-neonatal-pain?source=related\_link</a>
- 19 IASP (2011a). Acute Pain and Surgery. Global Year Against Acute Pain. [Online]. Tilgjengelig på

  <a href="http://www.iasp-pain.org/files/Content/ContentFolders/GlobalYearAgainstPain2/AcutePainFactSheets/7-Surgery.pdf">http://www.iasp-pain.org/files/Content/ContentFolders/GlobalYearAgainstPain2/AcutePainFactSheets/7-Surgery.pdf</a>
  [Lastet 14.april 2014].
- 20 Howard, R., Carter, B., Curry, J., Jain, A., Liossi, C., Morton, N., Rivett, K., Rose, M., Tyrrell, J., Walker, S., Williams, G. (2012). Good Practice in Postoperative and Procedural pain management. 2nd Edition. Pediatric Anesthesia, 22: 1–79. doi: 10.1111/j.1460-9592.2012.03838.x. <a href="http://onlinelibrary.wiley.com/doi/10.1111/j.1460-9592.2012.03838.x/epdf">http://onlinelibrary.wiley.com/doi/10.1111/j.1460-9592.2012.03838.x/epdf</a>
- 21 IASP (2011b). Interventions: Benefits and Barriers. Global Year Against Acute Pain. [Online]. Tilgjengelig på http://www.iasp-

Unique Protocol ID: 2014/7951

Secondary Ids: 2014/878 [Regional Committee for Medical Research Ethics Norway]

- pain.org/files/Content/ContentFolders/GlobalYearAgainstPain2/AcutePainFactSheets/2-Interventions.pdf [Lastet 14.april 2014].
- 22 Benhamou, D., Berti, M., Brodner, G., De Andres J, Draisci G, Moreno-Azcoita M, Neugebauer EA, Schwenk W, Torres LM, Viel E. (2007). Postoperative Analgesic THerapy Observational Survey (PATHOS): A practice pattern study in 7 Central/Southern Eurpean countries. *Pain*, 136, 134-141. <a href="http://www.sciencedirect.com/science/article/pii/S0304395907003545">http://www.sciencedirect.com/science/article/pii/S0304395907003545</a>
- 23 Reinertsen, H. (2008). Smerte hos barn. kap.3.I: Rustøen T & Wahl AK (red). *Ulike tekster om smerte fra nocisepsjon til livskvalitet*. Oslo, Gyldendal Norsk Forlag AS.
- 24 Smeland, A. & Reinertsen, H. (2012). Smertevurdering og behandling av postoperative smerter hos barn. *Tidsskriftet Kirurgen*, 1, 58-62. (5 s.). [Online]. Tilgjengelig på <a href="http://www.kirurgen.no/pdf/1201/">http://www.kirurgen.no/pdf/1201/</a> [Lastet 13.april 2014].
- 25 Bringuier S, Picot MC, Dadure C et al. (2009). A prospective comparison of post-surgical behavioral pain scales in preschoolers highlighting the risk of false evaluations. *Pain*, 145, 60-68.
- 26 Crelline, D., Sullivan, T. B., Babl, F. E., O'Sullivan, R., Hutchinson, A. (2007). Analysis of the validation of existing behavioral pain and distress scales for use in the procedural setting. *Pediatric Anesthesia*, 17, 720-733.
- 27 Ghai, B., Makkar. J.K. & Wig. J. (2008). Postoperative pain assessment in preverbal children and children with cognitive impairment. *Pediatric Anesthesia*, 18, 462-477.
- 28 Hicks, C.L., von Baeyer, C.L., Spafford, P. et al. (2001). The Faces Pain Scale-Revised: Toward a common metric in pain measurement. *Pain*, 93, 173-183.
- 29 Merkel, S.I., Voepel-Lewis, T. & Shayevitz et al. (1997). The FLACC: A Behavioral Scale for Scoring Postoperative Pain in Young Children. *Pediatric Nursing*, 23, 293-7.
- 30 Ellis, J. A., McCleary, L., Blouin, R., Dube, K., Rowley, B., MacNeil, M., & Cooke, C. (2007). Implementing best practice pain management in a pediatric hospital. *Journal for Specialists in Pediatric Nursing*, 12, 264-277. doi:10.1111/j.1744-6155.2007.00121.x
- 31 Johnston, C. C., Gagnon, A., Rennick, J., Rosmus, C., Patenaude, H., Ellis, J., Shapiro, C., Filion, F., Ritchie, J., Byron, J. (2007). One-on-one coaching to improve pain assessment and management practices of pediatric nurses. *Journal of Pediatric Nursing*, 22, 467-478. doi:10.1016/j.pedn.2007.07.004
- 32 Le May, S., Johnston, C. C., Choinière, M., Fortin, C., Kudirka, D., Murray, L., Chalut, D. (2009). Pain Management Practices in a Pediatric Emergency Room (PAMPER) Study: interventions with nurses. *Pediatr Emerg Care*. Aug;25(8):498-503. doi: 10.1097/PEC.0b013e3181b0a0af.
- 33 Vincent, C. V. H., Wilkie, D. J. & Wang, E. (2011). Pediatric Nurses' Beliefs and Pain Management Practices: An Intervention Pilot. *West J Nurs Res*, 33: 825 originally published online 20 December 2010
- 34 Björndal, A. & Hofoss, D. (2010). Statistikk for helse- og sosialfagene. (2 utg.). Oslo, Norge: Gyldendal Norsk Forlag AS.
- 35 Polit, D. & Beck, C. (2008). *Nursing research. Generating and Assessing Evidence for Nursing Practice*. Philadelphia, USA: Lippincott Williams & Williams.
- 36 Twycross, A., Finley, G. A. and Latimer, M. (2013). Pediatric nurses' postoperative pain management practices: An observational study. *Journal for Specialists in Pediatric Nursing*, 18: 189–201. doi: 10.1111/jspn.12026
- 37 Malterud, K. (2011). Kvalitative metoder i medisinsk forskning-en innføring. Oslo, Universitetssforlaget AS.
- 38 Kvale, S. & Brinkmann, S. (2010). Det kvalitative forskningsintervju. Oslo, Gyldendal Norsk Forlag AS.
- 39 Tjora, A. (2010). Kvalitative forskningsmetoder i praksis. Oslo: Gyldendal Norsk Forlag AS.
- 40 Williams, D. T., Wetton, N. and Moon, A. (1989). A Way In: Five Key Areas of Health Education. Health Education Authority, London.
- 41 Pridmore, P. & Bendelow, G. (1995) Images of health: exploring beliefs of children using the 'draw-and-write' technique. Health Education Journal, 54, 473–488.
- 42 Twycross, A., & Finley, G. A. (2013). Children's and parents' perceptions of postoperative pain management: a mixed methods study. *Journal of Clinical Nursing*, 22(21-22), 3095-3108. doi: 10.1111/jocn.12152 [Online]. Tilgjengelig på http://onlinelibrary.wiley.com/doi/10.1111/jocn.12152/pdf (13.04.2014).
- 43 Polkki T, Pietila AM, Vehvilainen-Julkunen K. (2003). Hospitalized children's descriptions of their experiences with postsurgical pain relieving methods. Int J Nurs Stud. Jan;40(1):33-44. PubMed PMID: 12550148. English.
- 44 Royal College of Nursing (2002). The Recognition and Assessment of Pain in Children: Audit Tool, RCN Publishing, London.
- 45 Creswell, JW (2009) Research Design: Qualitative, Quantitative, and Mixed Methods Approaches, Thousand Oaks: Sage.
- 46 Abdalrahim MS, Majali SA, Stomberg MW, <u>Bergbom I</u>. (2011). The effect of postoperative pain management program on improving nurses' knowledge and attitudes toward pain. <u>Nurse Educ Pract.</u>

Unique Protocol ID: 2014/7951

Secondary Ids: 2014/878 [Regional Committee for Medical Research Ethics Norway]

- 2011 Jul;11(4):250-5. doi: 10.1016/j.nepr.2010.11.016. Epub 2010 Dec 24. http://www.ncbi.nlm.nih.gov/pubmed/21186139
- 47 Forskningsetikkloven (2006). *Lov om behandling av etikk og redelighet i forskning* (Forskningsetikkloven). LOV 2006-06-30 nr 56. [Online]. Tilgjengelig på <a href="http://www.lovdata.no/all/hl-20060630-056.html">http://www.lovdata.no/all/hl-20060630-056.html</a> [Lastet 14.april 2014].
- 48 Helseforskningsloven (2008). *Lov om medisinsk og helsefaglig forskning* (Helseforskningsloven). LOV 2008-06-20 nr 44. [Online]. Tilgjengelig på <a href="http://www.lovdata.no/all/hl-20080620-044.html">http://www.lovdata.no/all/hl-20080620-044.html</a> [Lastet 14.april 2014].
- 49 Langtvedt, N. J. (2012). *Forskningsetikkloven*. De nasjonale forskningsetiske komiteer. [Online]. Tilgjengelig på <a href="http://www.etikkom.no/FBIB/Praktisk/Lover-og-retningslinjer/Forskningsetikkloven/">http://www.etikkom.no/FBIB/Praktisk/Lover-og-retningslinjer/Forskningsetikkloven/</a> [Lastet 14.april 2014].
- 50 Ruyter, K. W. (2009). *Medisin og helsefag*. De nasjonale forskningsetiske komiteer. Nedlastet fra http://www.etikkom.no/no/FBIB/Introduksjon/Innforing-i-forskningsetikk/Medisin-og-helsefag/
- 51 Fossheim, H., Hølen, J. & Ingierd, H. (2013). *Barn i forskningen etiske dimensjoner*. De nasjonale forskningsetiske komiteene. [Online]. Tilgjengelig på <a href="https://www.etikkom.no/Documents/Publikasjoner-som-PDF/Barn%20i%20forskning%20web.pdf">https://www.etikkom.no/Documents/Publikasjoner-som-PDF/Barn%20i%20forskning%20web.pdf</a>. [Lastet 14.april 2014].
- 52 Backe-Hansen, E. (2012). *Barn*. De nasjonale forskningsetiske komiteene. [Online]. Tilgjengelig på http://www.etikkom.no/FBIB/Temaer/Forskning-pa-bestemte-grupper/Barn/. [Lastet 14.april 2014].
- 53 Langtvedt, N. J. (2009). *Personvern*. De nasjonale forskningsetiske komiteer. [Online]. Tilgjengelig på <a href="http://www.etikkom.no/FBIB/Temaer/Personvern-og-ansvar-for-den-enkelte/Personvern/">http://www.etikkom.no/FBIB/Temaer/Personvern-og-ansvar-for-den-enkelte/Personvern/</a> [Lastet 14.april 2014].
- 54 Alver, B. G. (2009). *Ansvar for den enkelte*. (Sist oppdatert: 01. desember 2009). De nasjonale forskningsetiske komiteene. [Online]. Tilgjengelig på http://www.etikkom.no/FBIB/Temaer/Personvernog-ansvar-for-den-enkelte/Ansvar-for-den-enkelte/. [Lastet 14.april 2014].
- 55 Fossheim, H. J. (2009a). *Informert samtykke*. De nasjonale forskningsetiske komiteer. [Online]. Tilgjengelig på <a href="https://www.etikkom.no/FBIB/Temaer/Personvern-og-ansvar-for-den-enkelte/Informert-samtykke/">https://www.etikkom.no/FBIB/Temaer/Personvern-og-ansvar-for-den-enkelte/Informert-samtykke/</a> [Lastet 14.april 2014].
- 56 Norsk sykepleierforbund. (2011). Yrkesetiske retningslinjer for sykepleiere: ICNs etiske regler. Oslo: Norsk sykepleierforbund. [Online]. Tilgjengelig på <a href="https://www.sykepleierforbundet.no/ikbViewer/Content/785285/NSF-263428-v1-YER-hefte\_pdf.pdf">https://www.sykepleierforbundet.no/ikbViewer/Content/785285/NSF-263428-v1-YER-hefte\_pdf.pdf</a> [Lastet 14.april 2014].
- 57 Ruyter, K. W. (2000). Medisinsk forskningsetikk. I Ruyter, K. W., Førde, R. & J. H. Solbakk, J. H. *Medisinsk etikk en prblembasert tilnærming*. Gjøvik, Norge: Gyldendal Norsk Forlag AS.
- 58 Befring, E. (2010). Forskningsmetode med etikk og statistikk. (2 utg.). Fagernes: Valdres Trykkeri.
- 59 Fossheim, H. J. (2009b). *Konfidensialitet*. De nasjonale forskningsetiske komiteer. [Online]. Tilgjengelig på <a href="https://www.etikkom.no/FBIB/Temaer/Personvern-og-ansvar-for-den-enkelte/Konfidensialitet/">https://www.etikkom.no/FBIB/Temaer/Personvern-og-ansvar-for-den-enkelte/Konfidensialitet/</a> [Lastet 14.april 2014].
- 60 Langtvedt, N. J. (2009a). *Personopplysninger*. De nasjonale forskningsetiske komiteer. [Online]. Tilgjengelig på <a href="http://etikkom.no/no/FBIB/Temaer/Personvern-og-ansvar-for-den-enkelte/Personopplysninger/">http://etikkom.no/no/FBIB/Temaer/Personvern-og-ansvar-for-den-enkelte/Personopplysninger/</a> [Lastet 14.april 2014].
- 61 Langtvedt, N. J. (2009b). *Personvern*. De nasjonale forskningsetiske komiteer. [Online]. Tilgjengelig på <a href="http://etikkom.no/no/FBIB/Temaer/Personvern-og-ansvar-for-den-enkelte/Personvern/">http://etikkom.no/no/FBIB/Temaer/Personvern-og-ansvar-for-den-enkelte/Personvern/</a> [Lastet 14.april 2014].